CLINICAL TRIAL: NCT00688701
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter 12-week Study Assessing the Efficacy and Safety of AVE0010 in Patients With Type 2 Diabetes Not Treated With Antidiabetic Agents
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation in Monotherapy
Acronym: GETGOAL-MONO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC6018; EudraCT 2007-005887-29
Record Dates: First submitted 2008-05-07; First posted 2008-06-03 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia, GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Two-Step Titration) (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 12.
  Interventions: Drug: Placebo; Device: Pen auto-injector
- Placebo (One-Step Titration) (Placebo Comparator): 1-step initiation regimen of volume matching placebo: 10 mcg QD for 2 weeks, then 20 mcg QD up to Week 12.
  Interventions: Drug: Placebo; Device: Pen auto-injector
- Lixisenatide (Two-Step Titration) (Experimental): 2-step initiation regimen of lixisenatide: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 12.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector
- Lixisenatide (One-Step Titration) (Experimental): 1-step initiation regimen of lixisenatide: 10 mcg QD for 2 weeks, then 20 mcg QD up to Week 12.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide (One-Step Titration); Lixisenatide (Two-Step Titration)
Drug: Placebo — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo (One-Step Titration); Placebo (Two-Step Titration)
Device: Pen auto-injector
  Other Names: OptiClik®

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, used in a 2-step dose titration regimen in monotherapy, over a period of 12 weeks of treatment.

The primary objective is to assess the effects of lixisenatide, in comparison to placebo, on glycemic control using a 2-step dose titration regimen in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 12.

Secondary objectives are to assess the effects of lixisenatide, in comparison to placebo, on glycemic control in terms of HbA1c reduction when it is used in a one-step dose titration regimen over a period of 12 weeks, body weight, fasting plasma glucose (FPG), 2-hour postprandial plasma glucose (PPG) after a standardized meal, to assess the safety and tolerability, pharmacokinetics (PK) and anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, 4-arm, unbalanced design, parallel group study with a two-step titration regimen or a one-step titration regimen. The study is double-blind with regard to active and placebo treatments; however neither the study drug volume nor the titration regimens (that is, two-step or one-step) are blinded.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 2 months at the time of the screening visit, not treated with any antidiabetic agent

Exclusion Criteria:

* HbA1c less than (<) 7 percent (%) or greater than (>) 10%
* At the time of screening age < legal age of majority
* Pregnant or breastfeeding women and women of childbearing potential without effective contraceptive method of birth control
* Type 1 diabetes mellitus
* Type 2 diabetes treated by an antidiabetic agent within the 3 months preceding the study
* Fasting plasma glucose at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* Body mass index less than or equal to (<=) 20 kilogram per square meter (kg/m^2)
* Weight change of more than 5 kg during the previous 3 months
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within the previous year
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within the previous 3 months
* History of myocardial infarction, stroke, or heart failure requiring hospitalization within the previous 6 months
* Known history of drug or alcohol abuse within the previous 6 months
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension with a resting supine systolic or diastolic blood pressure >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase: >2 times the upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 ULN; total bilirubin: >1.5 ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter (g/dL) and/or neutrophils <1,500 per cubic mm (mm^3) and/or platelets <100,000/mm^3; positive test for Hepatitis B surface antigen and/or hepatitis C antibody
* Any clinically significant abnormality identified by physical examination, laboratory tests, electrocardiogram or vital sign at the time of screening that in the judgment of the investigator or any sub investigator precludes safe completion of the study or hinders the efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) within the previous 3 months
* Participation in any previous study with lixisenatide
* Use of any investigational drug within 3 months prior to study
* End-stage renal disease as defined by a calculated serum creatinine clearance of <15 milliliter/minute and/or patients on dialysis
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment, within the previous 6 months
* History of allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase: more than 2 injections missed; and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Tokyo, Japan
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- [Result] Fonseca VA, Alvarado-Ruiz R, Raccah D, Boka G, Miossec P, Gerich JE; EFC6018 GetGoal-Mono Study Investigators. Efficacy and safety of the once-daily GLP-1 receptor agonist lixisenatide in monotherapy: a randomized, double-blind, placebo-controlled trial in patients with type 2 diabetes (GetGoal-Mono). Diabetes Care. 2012 Jun;35(6):1225-31. doi: 10.2337/dc11-1935. Epub 2012 Mar 19. PMID 22432104
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 61 centers (68 were initiated) in 12 countries between May 14, 2008 and December 14, 2009.
Pre-assignment Details: A total of 795 patients were screened of which 434 (54.6%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 361 patients were randomized.
Groups:
- Placebo (Two-Step Titration): 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 12.
- Placebo (One-Step Titration): 1-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 2 weeks, then 20 mcg QD up to Week 12.
- Lixisenatide (Two-Step Titration): 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 12.
- Lixisenatide (One-Step Titration): 1-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 2 weeks, then 20 mcg QD up to Week 12.
Period: Overall Study
Arm/Group | Placebo (Two-Step Titration) | Placebo (One-Step Titration) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Started | 61 (Randomized) | 61 | 120 | 119
Treated/Safety Population | 61 (All patients who received at least 1 dose, regardless of amount of treatment administered.) | 61 | 120 | 119
Modified Intent-to-Treat(mITT)Population | 61 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 60 | 120 | 118
Subgroup for Standardized Meal Test | 27 (Patients at selected sites where standardized meal test was performed.) | 35 | 60 | 65
Completed | 57 | 56 | 110 | 108
Not Completed | 4 | 5 | 10 | 11
Not completed — Adverse Event | 1 | 0 | 5 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 8
Not completed — Poor compliance to protocol | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo (Combined): Included all patients who received 2-step initiation regimen of volume matching placebo and 1-step initiation regimen of volume matching placebo.
- Total: Total of all reporting groups
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration) | Total
Number analyzed (Participants) | 122 | 120 | 119 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.0) | 53.3 (9.7) | 53.8 (10.9) | 53.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 57 | 56 | 175
  Male | 60 | 63 | 63 | 186
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 90 | 88 | 85 | 263
  Race: Black | 3 | 0 | 3 | 6
  Race: Asian/Oriental | 24 | 27 | 29 | 80
  Race: Other | 5 | 5 | 2 | 12
  Ethnicity: Hispanic | 31 | 25 | 22 | 78
  Ethnicity: Non Hispanic | 91 | 95 | 97 | 283
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.07 (0.91) | 7.98 (0.92) | 8.07 (0.87) | 8.04 (0.90)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients analyzed = 60, 59 and 65 for Placebo (Combined), Lixisenatide (Two-Step Titration) and Lixisenatide (One-Step Titration) treatment arms, respectively, as meal challenge test was performed at selected sites only.
  mmol/L | 14.27 (4.84) | 14.81 (3.87) | 14.62 (3.41) | 14.57 (4.05)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 86.08 (22.21) | 89.04 (22.16) | 86.50 (21.00) | 87.20 (21.78)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 8.90 (2.16) | 9.15 (1.99) | 9.04 (1.97) | 9.03 (2.04)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients analyzed = 60, 59 and 65 for Placebo (Combined), Lixisenatide (Two-Step Titration) and Lixisenatide (One-Step Titration) treatment arms, respectively, as meal challenge test was performed at selected sites only.
  mmol/L | 4.82 (3.69) | 5.67 (3.05) | 5.34 (2.96) | 5.27 (3.25)
Duration of Diabetes [Median (Full Range); unit: years] | 1.37 [0.2 to 12.5] | 1.42 [0.2 to 21.5] | 1.11 [0.2 to 23.9] | 1.33 [0.2 to 23.9]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 31.76 (6.69) | 32.34 (6.72) | 31.65 (6.62) | 31.91 (6.66)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: Absolute change = HbA1c value at Week 12 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 12
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Lixisenatide (Two-Step Titration): 2-step initiation regimen of lixisenatide.
- Lixisenatide (One-Step Titration): 1-step initiation regimen of lixisenatide.
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 112 | 113 | 114
percentage of hemoglobin | -0.19 (0.121) | -0.73 (0.116) | -0.85 (0.119)
Statistical Analysis 1: Comparison: Placebo (Combined) vs Lixisenatide (Two-Step Titration); To detect a difference of 0.5% in change in HbA1c at Week 12 between 1 lixisenatide arm and placebo (combined), 120 patients per group would provide a power of 90% assuming common standard deviation of 1.2% with 2-sided test at 5% significance level. Statistical testing: 2-sided at significance level=0.05. Analysis of co-variance (ANCOVA) included treatment arms, randomization strata of screening HbA1c (<8.0,>=8.0%), BMI (<30,>=30 kg/m^2), country as fixed effects, baseline HbA1c as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Stepwise testing procedure applied to control type 1 error: Lixisenatide (2-step titration) was compared with Placebo (combined), if found statistically significant, then Lixisenatide (1-step titration) arm compared with Placebo (combined); Least squares (LS) mean difference = -0.54, 95% CI 2-sided [-0.785 to -0.300], Standard Error of Mean 0.123
Statistical Analysis 2: Comparison: Placebo (Combined) vs Lixisenatide (One-Step Titration); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.66, 95% CI 2-sided [-0.903 to -0.423], Standard Error of Mean 0.122

2. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) at Week 12
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal (performed in selected sites). Change was calculated by subtracting baseline value from Week 12 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 12
Population: Subgroup for standardized meal test. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 54 | 53 | 62
mmol/L | -0.65 (0.563) | -4.51 (0.572) | -5.47 (0.549)

3. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Description: Change was calculated by subtracting baseline value from Week 12 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 12
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 116 | 117 | 115
kilogram | -1.98 (0.341) | -1.96 (0.326) | -1.92 (0.338)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: Change was calculated by subtracting baseline value from Week 12 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 1 day after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 12
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 121 | 119 | 118
mmol/L | 0.19 (0.255) | -0.68 (0.247) | -0.89 (0.254)

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 12
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 12
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 112 | 113 | 114
percentage of participants | 26.8 | 52.2 | 46.5

6. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 12
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 112 | 113 | 114
percentage of participants | 12.5 | 31.9 | 25.4

7. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During the Double-Blind Treatment Period
Description: Routine fasting self monitored plasma glucose (SMPG) and central laboratory FPG values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG was performed. Threshold values for fasting SMPG/FPG: from baseline to Week 8: >270 milligram/deciliter (mg/dL) (15 mmol/L) and from Week 8 to Week 12: >240 mg/dL (13.3 mmol/L). For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 12
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 121 | 120 | 118
percentage of participants | 2.5 | 1.7 | 0.8

8. Other Pre Specified Outcome: Change From Baseline in Glucose Excursion at Week 12
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test (performed in selected sites), before study drug administration. Change was calculated by subtracting baseline value from Week 12 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 12
Population: Subgroup for standardized meal test. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 54 | 53 | 62
mmol/L | -0.67 (0.447) | -3.77 (0.454) | -4.36 (0.436)

9. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 12
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 116 | 117 | 115
percentage of participants | 17.2 | 16.2 | 18.3

10. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration)
Number analyzed (Participants) | 122 | 120 | 119
participants
  Symptomatic hypoglycemia | 2 | 3 | 1
  Severe symptomatic hypoglycemia | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration
Description: Median exposure to study treatment was 85 days for all treatment arms.The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo (Two-Step Titration): 2-step initiation regimen of volume matching placebo.
- Placebo (One-Step Titration): 1-step initiation regimen of volume matching placebo.
- Lixisenatide (Combined): Included all patients who received 2-step initiation regimen of lixisenatide and 1-step initiation regimen of lixisenatide.
Arm/Group | Placebo (Two-Step Titration) | Placebo (One-Step Titration) | Placebo (Combined) | Lixisenatide (Two-Step Titration) | Lixisenatide (One-Step Titration) | Lixisenatide (Combined)
Serious Adverse Events (participants affected / at risk) | 3/61 | 2/61 | 5/122 | 1/120 | 0/119 | 1/239
Other Adverse Events (participants affected / at risk) | 11/61 | 8/61 | 19/122 | 35/120 | 31/119 | 66/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Two-Step Titration) (N=61) | Placebo (One-Step Titration) (N=61) | Placebo (Combined) (N=122) | Lixisenatide (Two-Step Titration) (N=120) | Lixisenatide (One-Step Titration) (N=119) | Lixisenatide (Combined) (N=239)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Two-Step Titration) (N=61) | Placebo (One-Step Titration) (N=61) | Placebo (Combined) (N=122) | Lixisenatide (Two-Step Titration) (N=120) | Lixisenatide (One-Step Titration) (N=119) | Lixisenatide (Combined) (N=239)
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 9 | 4 | 13
Headache (Nervous system disorders) | 9 | 5 | 14 | 10 | 9 | 19
Nausea (Gastrointestinal disorders) | 3 | 2 | 5 | 29 | 24 | 53
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 8 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.